CLINICAL TRIAL: NCT04192396
Title: Prospective Study of the 'Win Test', a New Diagnostic Tool to Assess Human Endometrial Receptivity Under Natural Cycle or Hormone Replacement Therapy
Brief Title: Prospective Study of an Human Endometrial Receptivity Test
Acronym: Win-Test
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Merck Serono (GFI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0590
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Infertile
Keywords: Endometrial receptivity assessment for customized embryo transfer; Human Reproduction; ART; Endometrial receptivity
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RIF patients: Repeated implantation failure patients
- Oocyte/embryo donation program: Patients awaiting for oocyte/embryo-donation recipient patients

SUMMARY:
Evaluation of endometrial receptivity is a crucial step in in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) programs. Using "Omic technologies", such as transcriptomic and proteomic analyses, the investigators previously identified a specific molecular signature of human endometrial receptivity during the embryo implantation window. After validation of this signature in fertile women and in an ex vivo model (i.e., stromal and epithelial endometrium cells),the investigatorsdeveloped a diagnostic tool called Win-Test (Window Implantation Test) to evaluate the expression level of a set of endometrial receptivity-specific genes during the implantation window by quantitative RT-PCR. Based on their expression, each endometrial biopsy sample can be classified as receptive, partially receptive or non-receptive. Then, after the identification of the right cycle day within the implantation window where endometrium is considered as receptive, a customized timing for embryo transfer with respect of the synchronization of the embryo-maternal dialogue must be performed. A prospective study to validate the relevance of the Win-Test, is a necessary step to gauge its effectiveness. In this objective, patients with multiple implantation failures will be recruited. Embryo transfers were performed in double-arm: the intervention group had a customized timing of embryo transfer according to the Win-Test strategy and recommendation, the control group had their embryos transferred in a classical timing. Pregnancy and live birth rates (LBR) were compared between groups.

ELIGIBILITY:
Inclusion criteria :

* Infertile patients associated with multiple implantation failures.
* Signatures consent and non-opposition letter.
* Patients with a standard infertility assessment.
* Patients with a monitored cycle (ultrasound, hormonal markers) during the mock frozen embryo transfer cycle to perform the Win-test and during the embryo transfer cycle.
* Patients with complete treatment information during the mock frozen embryo transfer cycle to perform the Win-test and during the embryo transfer cycle.
* Patients with accurate transfer day information.
* Patients for whom we have the outcome (pregnancy, live birth).

Exclusion criteria:

More than 24 weeks of amenorrhea

Ages: 27 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women were recruited after written informed consent. All of them had a severe history of repeated implantation failures (RIFs). A classical infertility evaluation was performed including transvaginal sonography and uterine cavity was assessed by hysteroscopy. All patients were scheduled for replacement of cryopreserved embryos under hormone replacement therapy (HRT) or natural cycle. A mock frozen embryo transfer cycle, using a natural cycle or a HRT protocol, was monitored. Patients had endometrial biopsies performed through the presumed implantation window, 6 to 9 days after the LH (luteinizing hormone) surge for those on natural cycle or 5 to 9 days after the progesterone administration under HRT. Each biopsy was assessed for endometrial receptivity status using the Win-Test and assessment was stopped when appropriate endometrial receptivity was found. The clinical suitability of the Win-Test was performed in RIF patients who subsequently received Win-Test's guided embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | At 7-8 weeks of amenorrhea after customized timing of embryo transfer
  Clinical pregnancy was defined as ultrasound visualization of a gestational sac with a positive embryo heartbeat

SECONDARY OUTCOMES:
Live birth rate | More than 24 weeks of amenorrhea
  Live birth rate was defined as a delivery with at least one live born baby of more than 24 weeks of amenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Samir Hamamah, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Haouzi D, Entezami F, Torre A, Innocenti C, Antoine Y, Mauries C, Vincens C, Bringer-Deutsch S, Gala A, Ferrieres-Hoa A, Ohl J, Gonzalez Marti B, Brouillet S, Hamamah S. Customized Frozen Embryo Transfer after Identification of the Receptivity Window with a Transcriptomic Approach Improves the Implantation and Live Birth Rates in Patients with Repeated Implantation Failure. Reprod Sci. 2021 Jan;28(1):69-78. doi: 10.1007/s43032-020-00252-0. Epub 2020 Jul 28. PMID 32725589